CLINICAL TRIAL: NCT00668356
Title: PKPOP Study of Didanosine in HIV Treated Children, at Fasting Period and During the Meal
Brief Title: Bioequivalence Study of Didanosine in Children Treated for HIV
Acronym: ddI
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: questions of the benefit efficacy/risks of ddI during the meal not resolved
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Yannick VACHER, Department of Clinical Research of the Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P080101
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-01

CONDITIONS: HIV Infections
Keywords: HIV disease in children; HIV; children; didanosine; bioequivalence; pharmacokinetics; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Didanosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: didanosine
- 2 (Active Comparator)
  Interventions: Drug: didanosine

INTERVENTIONS:
Drug: didanosine — 28 days 400 mg/m2/day during the meal 28 days 240 mg/m2/day during fasting
  Arms: 2
Drug: didanosine — 28 days 240 mg/m2/day during fasting 28 days 400 mg/m2/day during the meal
  Arms: 1

SUMMARY:
The purpose of this study is to show that the administration of 400/mg/m2/day of didanosine(ddI) during the meal is bioequivalent to the administration of 240/mg/m2/day of didanosine during fasting, in HIV infected children treated by a ARV combination including ddI

DETAILED DESCRIPTION:
The didanosine is one of the reverse transcriptase inhibitors. This drug is efficient against the viral replication of the HIV. Licensing for the children was obtained in June, 1992. The main problem of the didanosine is its poor bioavailability: although gastro-resistant capsules were developed, its bioavailability remains dependent on alimentation. Taking a meal 1-2 hours before the administration of ddI leads to a reduction of 50% of its bioavailability as well for the child as for the adult. It is therefore recommended to take ddI during fasting period. This regimen in some cases can decrease therapeutic observance. A pharmacokinetic study of ddI will be conducted during the meal with 240 mg/m2/day during fasting period compare to 400 mg/m2/day during the meal. 26 patients, aged more than 6 years old, will be included and randomised in 2 groups. The first group will take the standard dose of ddI during 28 days during fasting period (phase A), then the high dose during the meal during 28 days (phase B). The second group will take first the phase B and secondly the phase A. Patients will be sequentially evaluated both after the first and the second period of treatment for pharmacokinetics and biological analysis.

ELIGIBILITY:
Inclusion Criteria:

* Children treated by the didanosine capsules more than 3 months
* viral load < 50 copies/ml
* written informed consent
* Normal renal function

Exclusion Criteria:

* Lack of observance
* Any treatments which can interact with ddI
* No written informed consent
* Weight > 60 kg

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
PK parameters | 28 days

SECONDARY OUTCOMES:
Biological analysis | 28 days
Quality of life | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Blanche, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Necker, Paris, France